CLINICAL TRIAL: NCT03561168
Title: Retrospective Review of Indications and Results of Brain MRI With Anesthesia/Sedation in Children Less Than Three Years of Age
Brief Title: Review of Diagnostic Yield of MRI Brain Results in Children Under Age 3 Years
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jamie Sinton, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-41288
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Seizures; Development Delay; Anesthetic Neurotoxicity
Keywords: Pediatric; MRI Indications; Anesthesia; Anesthetic Neurotoxicity; MRI Diagnostic Yield
MeSH Terms: conditions — Seizures; Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Developmental Delay: Children under age 3 who underwent MRI brain with anesthesia for the indication of Developmental Delay (between the dates of Dec 13, 2015 - Dec 13, 2016) at our institution.
  Interventions: Diagnostic Test: Change in plan of care based on MRI results
- Seizure: Children under age 3 who underwent MRI brain with anesthesia for the indication of Seizure (between the dates of Dec 13, 2015 - Dec 13, 2016) at our institution.
  Interventions: Diagnostic Test: Change in plan of care based on MRI results
- Developmental Delay and Seizure: Children under age 3 who underwent MRI brain with anesthesia for the indication of Developmental Delay and Seizure (between the dates of Dec 13, 2015 - Dec 13, 2016) at our institution.
  Interventions: Diagnostic Test: Change in plan of care based on MRI results

INTERVENTIONS:
Diagnostic Test: Change in plan of care based on MRI results — Study subjects have "received the intervention" if the results of their MRI either 1. provide an etiology for said MRI's indication or 2. the patient received a change in plan of care based on MRI results.

SUMMARY:
The investigators aim to identify the frequency with which an elective brain MRI yields and etiologic diagnosis to explain its indication. The protocol includes children undergoing elective brain MRI with anesthesia prior to their third birthday.

DETAILED DESCRIPTION:
On December 14, 2016 the FDA issued a warning regarding elective anesthetics in children under three years of age. While a single, short exposure to general anesthesia may not have negative effects on behavior or learning, repeated or prolonged anesthetics may affect brain development. To that end, minimizing exposure to elective general anesthetics if procedures are not clearly indicated in young children appeals to reason.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 0-36 months who received anesthesia (volatile gas anesthesia) or IV sedation (propofol, dexmedetomidine, barbiturates, benzodiazepines, or other agents) for brain MRI

Exclusion Criteria:

* MRI without sedation, brain MRI plus additional MRI imaging, i.e. spine, heart, etc., sedated MRI by a member of other department besides Anesthesiology.

Max Age: 1095 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under age 3 undergoing MRI brain with anesthesia or sedation between Dec 13, 2015 and Dec 13, 2016
Sampling Method: Non-Probability Sample
Enrollment: 561 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Etiologic diagnosis obtained from MRI brain | 1 year
  Determine the incidence of brain MRI abnormality that led to etiological explanation of developmental delay, autism or seizure.

SECONDARY OUTCOMES:
Quantify anesthetic exposure | 1 year
  To determine the doses of all anesthetic and sedative agents administered and the duration of anesthesia
Incidence of repeat MRI | 1 year
  To determine the incidence of repeat MRI scan in the study population. anesthesia. To determine the incidence of repeat MRI scan in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Dean B Andropoulos, MD, Study Director — Baylor College of Medicine; Jamie W Sinton, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a retrospective study, this question seems not applicable.

REFERENCES:
- [Background] Murias K, Moir A, Myers KA, Liu I, Wei XC. Systematic review of MRI findings in children with developmental delay or cognitive impairment. Brain Dev. 2017 Sep;39(8):644-655. doi: 10.1016/j.braindev.2017.04.006. Epub 2017 Apr 27. PMID 28457518
- [Background] Simpson GA, Colpe L, Greenspan S. Measuring functional developmental delay in infants and young children: prevalence rates from the NHIS-D. Paediatr Perinat Epidemiol. 2003 Jan;17(1):68-80. doi: 10.1046/j.1365-3016.2003.00459.x. PMID 12562474
- [Background] Rodriguez DP, Poussaint TY. Neuroimaging of the child with developmental delay. Top Magn Reson Imaging. 2007 Feb;18(1):75-92. doi: 10.1097/RMR.0b013e3180f63511. PMID 17607144
- [Background] Decobert F, Grabar S, Merzoug V, Kalifa G, Ponsot G, Adamsbaum C, des Portes V. Unexplained mental retardation: is brain MRI useful? Pediatr Radiol. 2005 Jun;35(6):587-96. doi: 10.1007/s00247-005-1406-x. Epub 2005 Mar 1. PMID 15739114
- [Background] Schaefer GB, Bodensteiner JB. Radiological findings in developmental delay. Semin Pediatr Neurol. 1998 Mar;5(1):33-8. doi: 10.1016/s1071-9091(98)80016-8. PMID 9548639
- [Background] Huang YY, Li L, Monteleone M, Ferrari L, States LJ, Riviello JJ, Kernie SG, Mencin AA, Gupta S, Sun LS. Use of Anesthesia for Imaging Studies and Interventional Procedures in Children. J Neurosurg Anesthesiol. 2016 Oct;28(4):400-404. doi: 10.1097/ANA.0000000000000355. PMID 27564559